CLINICAL TRIAL: NCT00248677
Title: Sensible Treatment of Obesity in Rural Youth
Brief Title: Sensible Treatment of Obesity in Rural Youth . . .
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK71555; R34DK071555 (NIH); 1R34DK071555-01 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

ARMS (3):
- No Contact Control (No Intervention)
- Behavior Family Intervention (Experimental)
  Interventions: Behavioral: Behavioral Family-Based Intervention
- Behavioral Parent-Only Intervention (Experimental)
  Interventions: Behavioral: Behavioral Parent-Based Intervention

INTERVENTIONS:
Behavioral: Behavioral Family-Based Intervention — Behavioral family intervention
  Arms: Behavior Family Intervention
Behavioral: Behavioral Parent-Based Intervention — Behavioral Parent-Only Intervention
  Arms: Behavioral Parent-Only Intervention

SUMMARY:
Project STORY (Sensible Treatment of Obesity in Rural Youth) will entail a three-arm randomized controlled trial to test the effectiveness of interventions designed to promote successful weight management in an important population, overweight children and their parents in medically underserved, rural settings. The current feasibility study will provide pilot data to develop and support a full-scale trial that will be implemented across multiple rural counties. In this pilot program, participants will be randomly assigned to one of two, 4-month long intervention programs that will be delivered in rural communities through Cooperative Extension Offices, or to a Wait List Control (WLC) group. The Behavioral Family-Based Intervention (BFI) will involve simultaneous, but separate treatment groups for both the child and their parent(s). The Behavioral Parent-Based Intervention (BPI) will involve groups for only the parent(s). Both programs will take a behavioral lifestyle approach to gradually modify dietary and physical activity patterns. The aims of the trial and its principal hypotheses are listed below.

AIMS:

* Evaluate the effects on child's standardized body mass index (BMI-z) of BPI and BFI delivered via group contacts to overweight children and/or their overweight parents in rural counties.
* Examine changes in children's dietary intake, physical activity, self-esteem, and body image.
* Compare the cost-effectiveness of the BPI and BFI.
* Evaluate the effects of the BPI and BFI on parent BMI.

DETAILED DESCRIPTION:
Project STORY (Sensible Treatment of Obesity in Rural Youth) will entail a three-arm randomized controlled trial to test the effectiveness of interventions designed to promote successful weight management in an important population, overweight children and their parents in medically underserved, rural settings. The current feasibility study will provide pilot data to develop and support a full-scale trial that will be implemented across multiple rural counties. In this pilot program, participants will be randomly assigned to one of two, 4-month long intervention programs that will be delivered in rural communities through Cooperative Extension Offices, or to a Wait List Control (WLC) group. The Behavioral Family-Based Intervention (BFI) will involve simultaneous, but separate treatment groups for both the child and their parent(s). The Behavioral Parent-Based Intervention (BPI) will involve groups for only the parent(s). Both programs will take a behavioral lifestyle approach to gradually modify dietary and physical activity patterns. The aims of the trial and its principal hypotheses are listed below.

AIMS:

* Evaluate the effects on child's standardized body mass index (BMI-z) of BPI and BFI delivered via group contacts to overweight children and/or their overweight parents in rural counties.
* Examine changes in children's dietary intake, physical activity, self-esteem, and body image.
* Compare the cost-effectiveness of the BPI and BFI.
* Evaluate the effects of the BPI and BFI on parent BMI.

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: all ethnic groups.
* Sex/Gender of Child Participant: Males and females.
* Age of Child Participant: 8 - 12 years.
* Child's Body-Mass Index: BMI above the 85th percentile for sex and age.
* Participating Parent or Legal Guardian: Must have participating parent or legal guardian (male or female) with BMI > 25 kg/m2. Participants (children and parents) must weigh less than 159 kg (350 pounds) in order to allow weight measurement on a standard balance beam scale.
* Physician Authorization: Letter signed by a physician medically clearing individuals (children and adults) to participate in weight management program. For families who are not able to access physician care, we will arrange for an appointment with a health care provider.
* Place of Residence: Child and participating parents must live in a rural county and within the same house.

Exclusion Criteria:

* Child or participating parent has dietary or exercise restrictions, or a medical condition that contraindicates mild energy restriction or moderate physical activity: history of musculo-skeletal condition that limits walking; heart condition; diabetes; chronic lung diseases limiting physical activity; uncontrolled high blood pressure or uncontrolled exercise induced-asthma as determined by a physician.
* Participating parent pregnant or plans on becoming pregnant within the next year.
* Medication exclusions: Child or participating parent on antipsychotic agents; systemic corticosteroids; or current use of prescription weight-loss drugs, insulin, or other diabetic medications.
* Child or participating parent currently engaged in another weight control program.
* Conditions or behaviors likely to affect the conduct of the trial: unwilling or unable to give informed consent; parent or legal guardian unable to read English at the 5th grade level; unwilling to accept random assignment; unable to travel to extension office for intervention sessions; likely to move out of the county within the next 18 months; child or parent with major psychiatric disorder; child with major cognitive or developmental delay; children with a current pattern of aggressive or oppositional behavior; or any other condition/situation which in the opinion of staff would adversely affect participation in Project STORY.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in Child BMI Z-score | Sept 2005 - Aug 2008

SECONDARY OUTCOMES:
Change in parent BMI | Sept 2005 - Aug 2008
Change in child dietary intake | Sept 2005 - Aug 2008
Change in child's physical activity and steps per day | Sept 2005 - Aug 2008

CONTACTS AND LOCATIONS:
Overall Officials: David M. Janicke, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States